CLINICAL TRIAL: NCT04204616
Title: A Prospective, Multicenter, Long-Term Study to Assess the Safety and Efficacy of Nemolizumab (CD14152) in Subjects With Prurigo Nodularis
Brief Title: A Long-term Study of Nemolizumab (CD14152) in Participants With Prurigo Nodularis (PN)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.202699; 2019-004294-13 (EudraCT Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — nemolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nemolizumab (Experimental): Participants weighing less than (<) 90kilogram (kg) will receive 30 milligram (mg) nemolizumab every 4 weeks (Q4W) and participants weighing greater than or equal to (>=) 90 kg will receive 60 mg nemolizumab (two 30-mg injections) Q4W.
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Nemolizumab — Nemolizumab 30 mg will be administered as subcutaneous (SC) injection.
  Other Names: CD14152

SUMMARY:
The primary purpose of this study is to assess the long-term safety of nemolizumab (CD14152) in participants with prurigo nodularis (PN).

ELIGIBILITY:
Inclusion Criteria:

* Participants who may benefit from study participation in the opinion of the investigator and participated in a prior nemolizumab study for PN including: (a). Participants who completed the treatment period in a phase 3 pivotal study (NCT04501666 or NCT04501679) and enroll within 56 days OR (b). Participants who were previously randomized in the nemolizumab phase 2a PN study (NCT03181503) OR (c). Participants who completed through Week 24 of the phase 3b durability study (NCT05052983) or who exit the study due to relapse may be eligible to re-enter in the LTE study within 28 days of exiting the durability study (selected countries/ selected sites)
* Female participants of childbearing potential (that is, fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree either to be strictly abstinent throughout the study and for 12 weeks after the last study drug injection, or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection
* Participant willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol, including periodic weekly recordings by the participant using an electronic handheld device provided for this study
* Understand and sign an informed consent form (ICF) before any investigational procedure(s) are performed

Exclusion Criteria:

* Participants who, during their participation in a prior nemolizumab study, experienced an adverse event (AE) which in the opinion of the investigator could indicate that continued treatment with nemolizumab may present an unreasonable risk for the participant
* Body weight < 30 kg
* Pregnant women (positive pregnancy test result at screening or baseline visit or re-entry Week R0 visit), breastfeeding women, or women planning a pregnancy during the clinical study
* Any medical or psychological condition that may put the participant at significant risk according to the investigator's judgment, if he/she participates in the clinical study, or may interfere with study assessments (example, poor venous access or needle-phobia)
* Planning or expected to have a major surgical procedure during the clinical study
* Participants unwilling to refrain from using prohibited medications during the clinical study
* History of alcohol or substance abuse within 6 months prior to the screening visit or re-entry Week R0 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) by Severity | Up to 192 weeks
  Incidence of AEs including AEs of Special Interest (AESIs), Treatment Emergent AEs (TEAEs) and Serious AEs (SAEs) by severity as mild, moderate or severe will be reported. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with relevant investigational product. SAE is any untoward medical occurrence that at any dose may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. TEAE is an AE that occurs on or after the first date of study drug(s) administration until the date of last study visit. An AESI is a noteworthy treatment-emergent event for the study drug that should be monitored closely and reported promptly.

SECONDARY OUTCOMES:
Percentage of Participants with an Investigator Global Assessment (IGA) Success up to Week 184 | Up to Week 184
  Percentage of participants with an IGA success (defined as IGA of 0 [Clear] or 1 [Almost clear]) up to Week 184 will be reported.
Percentage of Participants with an Improvement of >=4 from Baseline in Peak Pruritus (PP) Numeric Rating Scale (NRS) up to Week 184 | Baseline up to Week 184
  Percentage of participants with an improvement of >= 4 from baseline in PP NRS up to Week 184 will be reported. The PP NRS has a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percentage of Participants with Low Disease Activity State up to Week 184 | Up to Week 184
  Percentage of participants with low disease activity state (that is, IGA less than or equal to [<=]2) up to Week 184 will be reported.
Percentage of Pruriginous Lesions with Excoriations/Crusts up (PAS item 5a) up to Week 184 | Up to Week 184
  Prurigo Activity Score (PAS) will include a count of the number of lesions in a representative area and a calculated staging (stage 0 to stage 4) based on the percentage of lesions with excoriations/crusts and healed lesions compared to all lesions. PAS item 5a reflects the current itch/scratch activity. It is used to estimate what percentage of the pruriginous legions show excoriations/crusts. 100 percent (%) = All pruriginous lesions have excoriations/crusts. Percentage of pruriginous lesions with excoriations/crusts (PAS item 5a) up to Week 184 will be reported.
Percentage of Healed Prurigo Lesions (PAS item 5b) up to Week 184 | Up to Week 184
  PAS item 5b item reflects the stage of the prurigo. It is used to estimate what percentage of the pruriginous lesions have healed.100% = all pruriginous lesions have healed. Percentage of healed prurigo lesions (PAS item 5b) up to Week 184 will be reported.
Change from Baseline in Number of Lesions in Representative Area (PAS item 4) up to Week 184 | Baseline up to Week 184
  Change from baseline in number of lesions in representative area (PAS item 4) up to Week 184 will be reported.
Percentage of Participants with PP NRS <2 up to Week 184 | Up to Week 184
  Percentage of participants with PP NRS <2 up to Week 184 will be reported. PP NRS is a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percent Change from Baseline in PP NRS up to Week 184 | Baseline up to Week 184
  Percent change from baseline in PP NRS up to Week 184 will be reported. PP NRS is a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Absolute Change from Baseline in PP NRS up to Week 184 | Baseline up to Week 184
  Absolute change from baseline in PP NRS up to Week 184 will be reported. PP NRS is a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percentage of Participants with Average Pruritus (AP) NRS <2 up to Week 52 | Up to Week 52
  Percentage of participants with AP NRS less than (<) 2 up to Week 52 will be reported. AP NRS has a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percentage of Participants with an Improvement of >=4 from Baseline in AP NRS up to Week 52 | Up to Week 52
  Percentage of participants with an improvement of >=4 from baseline in AP NRS up to Week 52 will be reported. AP NRS has a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percent Change from Baseline in AP NRS up to Week 52 | Up to Week 52
  Percent change from baseline in AP NRS up to Week 52 will be reported. AP NRS has a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Absolute Change from Baseline in AP NRS up to Week 52 | Up to Week 52
  Absolute change from baseline in AP NRS up to Week 52 will be reported. AP NRS has a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Percentage of Participants with an Improvement of >=4 from Baseline in Sleep Disturbance (SD) NRS up to Week 184 | Up to Week 184
  Percentage of participants with an improvement of >=4 from baseline in Sleep Disturbance (SD) NRS up to Week 184 will be reported. SD NRS has a scale of 0 to 10, with 0 being "no sleep loss related to the symptoms of my skin disease (prurigo nodularis)" and 10 being "I did not sleep at all due to the symptoms of my skin disease (prurigo nodularis)".
Percent Change from Baseline in SD NRS up to Week 184 | Up to Week 184
  Percent change from baseline in SD NRS up to Week 184 will be reported. SD NRS has a scale of 0 to 10, with 0 being "no sleep loss related to the symptoms of my skin disease (prurigo nodularis)" and 10 being "I did not sleep at all due to the symptoms of my skin disease (prurigo nodularis)".
Absolute Change from Baseline in SD NRS up to Week 184 | Up to Week 184
  Absolute change from baseline in SD NRS up to Week 184 will be reported. SD NRS has a scale of 0 to 10, with 0 being "no sleep loss related to the symptoms of my skin disease (prurigo nodularis)" and 10 being "I did not sleep at all due to the symptoms of my skin disease (prurigo nodularis)".
Change from Baseline in Prurigo Nodularis (PN)-associated Pain Frequency up to Week 184 | Baseline up to Week 184
  Change from baseline in PN-associated pain frequency up to Week 184 will be reported. The pain frequency will be assessed on a scale of 0 to 5 where 0 = never, 1 = less than once a week, 2 = 1-2 days a week, 3 = 3-4 days a week, and 4 = 5-6 days a week.
Change from Baseline in PN-associated Pain Intensity up to Week 184 | Baseline up to Week 184
  Change from baseline in PN-associated pain intensity up to Week 184 will be reported. The pain intensity will be assessed on a scale of 0 to 10, with 0 being "no pain" and 10 being "the worst unbearable pain".
Percentage of Participants Reporting low Disease Activity Based on Patient Global Assessment of Disease (PGAD) up to Week 52 | Up to Week 52
  Percentage of participants reporting low disease activity (clear, almost clear, or mild) based on Patient Global Assessment of Disease (PGAD) up to Week 52 to be reported.
Percentage of Participants Satisfied with Study Treatment Based on Patient Global Assessment of Treatment (PGAT) up to Week 52 | Up to Week 52
  Percentage of participants satisfied with study treatment (good, very good, or excellent) based on Patient Global Assessment of Treatment (PGAT) up to Week 52 will be reported.
Percentage of Participants with a Change of >=4 from Baseline in Dermatology Life Quality Index (DLQI) up to Week 184 | Baseline up to Week 184
  Percentage of participants with a change of >=4 from baseline in Dermatology Life Quality Index (DLQI) up to Week 184 will be reported. The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily activities, leisure, work/school, personal relationships, and treatment. The participant will rate each question ranging from 0 (not at all) to 3 (very much). A higher total score indicates a poorer quality of life (QoL).
Change from Baseline in EuroQoL 5-Dimension (EQ-5D) up to Week 184 | Baseline up to Week 184
  Change from baseline in EuroQoL 5-Dimension (EQ-5D) up to Week 184 will be reported. The EQ-5D instrument is a validated questionnaire, completed by the participant that consists of 2 parts. The first part consists of 5 multiple choice QoL questions and the second is a 100 point Visual Analog Scale (VAS) with 0 being "Worst imaginable health state" and 100 being "Best imaginable health state".
Time to Permanent Study Drug Discontinuation | Baseline to 184 weeks
Time to Rescue Therapy | Baseline to 184 weeks
Percentage of Participants Receiving Any Rescue Treatment by Rescue Treatment | Baseline up to 184 weeks

CONTACTS AND LOCATIONS:
Locations (147):
- United States (54):
  - Galderma Investigational Site, Birmingham, Alabama
  - Galderma Investigational Site, Fountain Valley, California
  - Galderma Investigational Site, Los Angeles, California
  - Galderma Investigational Site, San Diego, California
  - Galderma Investigational Site, Santa Monica, California
  - Galderma Investigational Site, Washington D.C., District of Columbia
  - Galderma Investigational Site, Aventura, Florida
  - Galderma Investigational Site, Delray Beach, Florida
  - Galderma Investigational Site, Hollywood, Florida
  - Galderma Investigational Site, Largo, Florida
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, North Miami Beach, Florida
  - Galderma Investigational Site, Ormond Beach, Florida
  - Galderma Investigational Site, Pembroke Pines, Florida
  - Galderma Investigational Site, Tampa, Florida
  - Galderma Investigational Galderma Investigational Site, Columbus, Georgia
  - Galderma Investigational Site, Macon, Georgia
  - Galderma Investigational Site, Newnan, Georgia
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Galderma Investigational Site, Chicago, Illinois
  - Galderma I Galderma Investigational Site, Lake Bluff, Illinois
  - Galderma Investigational Site, Indianapolis, Indiana
  - Galderma Investigational Site, Topeka, Kansas
  - Galderma Investigational Site, Louisville, Kentucky
  - Galderma Investigational Site, Baltimore, Maryland
  - Galderma Investigational Site, Boston, Massachusetts
  - Galderma Investigational Site, Ann Arbor, Michigan
  - Galderma Investigational Site, Saint Joseph, Michigan
  - Galderma Investigational Site, Saint Joseph, Missouri
  - Galderma Investigational Site, St Louis, Missouri
  - Galderma Investigational Site, Henderson, Nevada
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational Galderma Investigational Site, New York, New York
  - Galderma Investigational Site, High Point, North Carolina
  - Galderma Investigational Site, Raleigh, North Carolina
  - Galderma Investigational Site, Winston-Salem, North Carolina
  - Galderma Investigational Site, Cincinnati, Ohio
  - Galderma Investigational Site, Cleveland, Ohio
  - Galderma Investigational Site, Dublin, Ohio
  - Galderma Investigational Site, Philadelphia, Pennsylvania
  - Galderma Investigational Site, Anderson, South Carolina
  - Galderma Investigational Site, Knoxville, Tennessee
  - Galderma Investigational Site, Murfreesboro, Tennessee
  - Galderma Investigational Galderma Investigational Site, Austin, Texas
  - Galderma Investigational Site, Dallas, Texas
  - Galderma Investigational Site, Dripping Springs, Texas
  - Galderma Investigational Site, Houston, Texas
  - Galderma Investigational Site, Pflugerville, Texas
  - Galderma Investigational Site, Webster, Texas
  - Galderma Investigational Site, Salt Lake City, Utah
  - Galderma Investigational Galderma Investigational Site, Springville, Utah
  - Galderma Investigational Site, Fairfax, Virginia
  - Galderma Investigational Site, Lynchburg, Virginia
  - Galderma Investigational Site, Morgantown, West Virginia
- Austria (3):
  - Galderma Investigational Site, Graz
  - Galderma Investigational Site, Linz
  - Galderma Investigational Site, Vienna
- Belgium (5):
  - Galderma Investigational Site, Brussels
  - Galderma Investigational Site, Ghent
  - Galderma Investigational Site, Jette
  - Galderma Investigational Site, Leuven
  - Galderma Investigational Site, Liège
- Canada (8):
  - Galderma Investigational Site, Calgary, AL
  - Galderma Investigational Site, London, Ontario
  - Galderma Investigational Site, North York, Ontario
  - Galderma Investigational Site, Saskatoon, Saskatchewan
  - Galderma Investigational Site, Calgary
  - Galderma Investigational Site, London
  - Galderma Investigational Site, Markham
  - Galderma Investigational Site, Toronto
- Denmark (2):
  - Galderma Investigational Site, Aarhus
  - Galderma Investigational Site, Hellerup
- France (10):
  - Galderma Investigational Site, Bordeaux
  - Galderma Investigational Site, Brest
  - Galderma Investigational Site, Nantes
  - Galderma Investigational Site, Nice
  - Galderma Investigational Site, Paris
  - Galderma Investigational Site, Pierre-Bénite
  - Galderma Investigational Site, Rouen
  - Galderma Investigational Site, Saint-Etienne
  - Galderma Investigational Site, Toulouse
  - Galderma Investigational Site, Valence
- Germany (19):
  - Galderma Investigational Site, Aachen
  - Galderma Investigational Site, Augsburg
  - Galderma Investigational Site, Bad Bentheim
  - Galderme Investigational Site, Berlin
  - Galderma Investigational Site, Bonn
  - Galderma Investigational Site, Darmstadt
  - Galderma Investigational Site, Dresden
  - Galderma Investigational Site, Düsseldorf
  - Galderma Investigational Site, Eppendorf
  - Galderma Investigational Site, Göttingen
  - Galderma Investigational Site, Halle
  - Galderma Investigational Site, Hamburg
  - Galderma Investigational Site, Heidelberg
  - Galderma Investigational Site, Kiel
  - Galderma Investigational Site, Lübeck
  - Galderma Investigational Site, Mainz
  - Galderma Investigational Site, Münich
  - Galderma Investigational Site, Münster
  - Galderma Investigational Site, Tübingen
- Hungary (3):
  - Galderma Investigational Site, Kecskemét
  - Galderma Investigational Site, Szeged
  - Galderma Investigational Site, Szolnok
- Italy (10):
  - Galderma Investigational Site, Catania
  - Galderma Investigational Site, Chieti
  - Galderma Investigational Site, Genova
  - Galderma Investigational Site, L’Aquila
  - Galderma Investigational Site, Modena
  - Galderma Investigational Site, Napoli
  - Galderma Investigational Site, Parma
  - Galderma Investigational Site, Perugia
  - Galderma Investigational Site, Roma
  - Galderma Investigational Site, Vicenza
- Netherlands (2):
  - Galderma Investigational Site, Groningen
  - Galderma Investigational Site, Utrecht
- Poland (16):
  - Galderma Investigational Site, Bydgoszcz
  - Galderma Investigational Site, Chorzów
  - Galderma Investigational Site, Częstochowa
  - Galderma Investigational Site, Gdansk
  - Galderma Investigational Site, Gdynia
  - Galderma Investigational Site, Katowice
  - Galderma Investigational Site, Krakow
  - Galderma Investigational Site, Lodz
  - Galderma Investigational Site, Lublin
  - Galderma Investigational Site, Olsztyn
  - Galderma Investigational Site, Ostrowiec Świętokrzyski
  - Galderma Investigational Site, Poznan
  - Galderma Investigational Site, Rzeszów
  - Galderma Investigational Site, Szczecin
  - Galderma Investigational Site, Warsaw
  - Galderma Investigational Site, Wroclaw
- South Korea (2):
  - Galderma Investigational Site, Gyeonggi-do
  - Galderma Investigational Site, Seoul
- Spain (2):
  - Galderma Investigational Site, Barcelona
  - Galderma Investigational Site, Las Palmas de Gran Canaria
- Galderma Investigational Site, Solna, Sweden
- Switzerland (6):
  - Galderma Investigational Site, Bern
  - Galderma Investigational Site, Buochs
  - Galderma Investigational Site, Lausanne
  - Galderma Investigational Site, Obbürgen
  - Galderma Investigational Site, Sankt Gallen
  - Galderma Investigational Site, Weinfelden
- United Kingdom (4):
  - Galderma Investigational Site, Dudley
  - Galderma Investigational Site, Glasgow
  - Galderma Investigational Site, London
  - Galderma Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Legat FJ, Kwatra SG, Reich A, Boulinguez S, Tsianakas A, Sauder M, Barbarot S, Szepietowski JC, Conrad C, Pink AE, Weisshaar E, Misery L, Metz M, Laquer VT, Sivamani RK, Yosipovitch G, Thaci D, Skov L, Chen X, Noda A, Jabbar-Lopez ZK, Piketty C, Stander S. Nemolizumab in prurigo nodularis up to 100 weeks: OLYMPIA LTE interim analysis. J Eur Acad Dermatol Venereol. 2025 Dec 17. doi: 10.1111/jdv.70266. Online ahead of print. PMID 41405008